CLINICAL TRIAL: NCT01380756
Title: A Phase 1 Study Evaluating the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Orally Administered AMG 900 in Adult Subjects With Acute Myeloid Leukemia
Brief Title: Study Evaluating Orally Administered AMG 900 in Adult Subjects With Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20101351
Record Dates: First submitted 2011-06-09; First posted 2011-06-27 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Cancer; Hematologic Malignancies; Leukemia; Myeloid Leukemia
Keywords: Amgen; Phase 1; Clinical Trial; Aurora kinase inhibitor; Open label; Oncology; Hematology
MeSH Terms: conditions — Neoplasms; Hematologic Neoplasms; Leukemia; Leukemia, Myeloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1- Dose Escalation (Experimental): The dose escalation will be conducted in 2 parts. Group 1 will consist of 8 cohorts and Group 2 will consist of 5 cohorts. The dose escalation is aimed at determining the maximum tolerated dose (MTD) of AMG 900.
  Interventions: Drug: Arm 1- Dose Escalation
- Arm 2- Dose Expansion (Experimental): The dose expansion part of the study will begin after completion of the dose escalation phase and will consist of 20 subjects with acute myelogenous leukemia.
  Interventions: Drug: Arm 2- Dose Expansion

INTERVENTIONS:
Drug: Arm 1- Dose Escalation — AMG 900 is a small molecule aurora kinase inhibitor. AMG 900 will be administered daily for 4 days every 2 weeks or daily 7 days every 2 weeks (ie.g., 4 consecutive days of dosing followed by 10 consecutive days off treatment).
  Arms: Arm 1- Dose Escalation
Drug: Arm 2- Dose Expansion — AMG 900 is a small molecule aurora kinases inhibitor. The dose expansion phase would be conducted to gain further clinical experience with AMG 900 in AML at the optimal dose schedule.
  Arms: Arm 2- Dose Expansion

SUMMARY:
This study of AMG 900 will be conducted in two parts: dose escalation and dose expansion. The dose escalation part of the study is aimed at evaluating the safety, tolerability and PK (pharmacokinetics) of oral AMG 900 in subjects with acute myeloid leukemia. Up to 93 subjects may be enrolled in dose escalation. The dose expansion part of the study will consist of 20 subjects with acute myeloid leukemia. The dose of AMG 900 will be dependent upon data from the dose escalation part of the study.

ELIGIBILITY:
Inclusion Criteria:

* Men or women ≥ 18 years old
* Pathologically documented, definitively diagnosed AML that has failed standard treatments or for which no standard therapy is available or the subject refuses standard therapy
* Must consent to undergo bone marrow biopsies per schedule of assessments

Exclusion Criteria:

* White blood cell greater than 20,000 uL
* History of or active central nervous system leukemia
* Prior allogeneic bone marrow transplant
* Subject will not be available for protocol-required study visits or procedures

Other Inclusion/ Exclusion Criteria may apply to qualify for enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2011-10-04 (Actual); Primary Completion 2014-09-04 (Actual); Study Completion 2014-09-04 (Actual)

PRIMARY OUTCOMES:
Subject incidence of adverse events | 1 year
Subject incidence of dose limiting toxicities (DLTs) | 1 year
Maximum observed concentration of AMG 900 | 1 year
Time to maximum observed concentration of AMG 900 | 1 year
Area under the plasma concentration-time curve (AUC) of AMG 900 | 1 year
Half life of AMG 900 | 1 year

SECONDARY OUTCOMES:
Objective response as per Cheson Response Criteria | 1 year
Change in the number of p-Histone H3 positive cells from baseline | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (3):
- United States (3):
  - Research Site, Stony Brook, New York
  - Research Site, Cleveland, Ohio
  - Research Site, Houston, Texas

REFERENCES:
- [Background] Kantarjian HM, Schuster MW, Jain N, Advani A, Jabbour E, Gamelin E, Rasmussen E, Juan G, Anderson A, Chow VF, Friberg G, Vogl FD, Sekeres MA. A phase 1 study of AMG 900, an orally administered pan-aurora kinase inhibitor, in adult patients with acute myeloid leukemia. Am J Hematol. 2017 Jul;92(7):660-667. doi: 10.1002/ajh.24736. Epub 2017 Jun 5. PMID 28370201
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com